CLINICAL TRIAL: NCT04983719
Title: Fertility-sparing Management of a Suspicion of Leiomyosarcoma: Avoiding Hysterectomy by Performing Transcervical Myoma Biopsy
Brief Title: Transcervical Myoma Biopsy Video
Acronym: TMBV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0496
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Atypical; Myoma
Keywords: YOUNG WOMAN WITH DESIRE FOR PREGNANCY; ATYPICAL MYOMA; FERTILITY PRESERVATION; BIOPSY
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the fertility-sparing management of an atypical uterine myoma. Step-by-step video explanation of transcervical biopsy using transabdominal ultrasound guidance, highlighting tips and tricks. Patient consent was obtained for publication of the case.

ELIGIBILITY:
Inclusion criteria:

* age >18 years old
* WOMAN WITH DESIRE FOR PREGNANCY
* ATYPICAL MYOMA

Exclusion criteria:

- age < 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: YOUNG WOMAN WITH DESIRE FOR PREGNANCY AND ATYPICAL MYOMA
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of video | day 1
  BIOPSY TECHNIQUE DESCRIBED BY VIDEO

CONTACTS AND LOCATIONS:
Overall Officials: GAUTHIER RATHAT, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC